CLINICAL TRIAL: NCT04112823
Title: Dexamethasone for Acute Migraine. A Randomized Dose-comparison Study
Brief Title: Dexamethasone for Migraine - Dose Comparison
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-10562
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone 4mg (Active Comparator): Dexamethasone 4mg, administered intravenously
  Interventions: Drug: Dexamethasone 4mg
- Dexamethasone 16mg (Active Comparator): Dexamethasone 16mg, administered intravenously
  Interventions: Drug: Dexamethasone 16mg

INTERVENTIONS:
Drug: Dexamethasone 4mg — Dexamethasone 4mg + metoclopramide 10mg, intravenously
  Other Names: Dexasone 4 mg
  Arms: Dexamethasone 4mg
Drug: Dexamethasone 16mg — Dexamethasone 16mg + metoclopramide 10mg, intravenously
  Other Names: Dexasone 16 mg
  Arms: Dexamethasone 16mg

SUMMARY:
Dexamethasone is an evidence-based treatment of acute migraine. This is a randomized comparison of two different doses of dexamethasone for acute migraine.

All patients will also be treated with metoclopramide.

DETAILED DESCRIPTION:
Investigational medications. Medications in each study arm are as follows:

A. Metoclopramide 10mg IV drip over 15 minutes (for acute treatment)+ dexamethasone 4 mg IV B. Metoclopramide 10mg IV drip over 15 minutes (for acute treatment)+ dexamethasone 16 mg IV Assignment. Will be concealed. The research pharmacist will determine assignment based on a random number sequence. Randomization. Randomization will occur in blocks of 4 based on a random number generator. Blinding. Patients, clinicians, and research personnel will be blinded. Stratification. Subjects will be stratified by study site (Moses or Weiler) and baseline pain intensity (moderate or severe).

Follow-up phone calls will be performed 48 hours and 7 days after ED (emergency department) discharge. At the first call, the next follow-up phone call will be scheduled. Attempts to complete the follow-up calls successfully will be made every eight hours until deemed futile. At this point, questionnaires will be sent by express courier, and failing this, the investigator will perform a home visit.

At the 48-hour phone call, the focus will be assessments of pain, functional status, migraine associated features, adverse events, satisfaction with the medication received, and use of rescue medication. The focus of the seven day phone call will be on the total number of days with headache since ED discharge, the need for repeat ED visits, healthcare providers visited, days of work missed, and adverse medication effects.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe migraine

Exclusion Criteria:

* Medication contra-indication
* Concern for secondary cause of headache

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 209 (Actual)
Dates: Start 2019-12-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedman BW, Solorzano C, Kessler BD, Martorello K, Lutz CL, Feliciano C, Adler N, Moss H, Cain D, Irizarry E. Randomized Trial Comparing Low- vs High-Dose IV Dexamethasone for Patients With Moderate to Severe Migraine. Neurology. 2023 Oct 3;101(14):e1448-e1454. doi: 10.1212/WNL.0000000000207648. Epub 2023 Aug 21. PMID 37604662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced in December 2019, was paused between March and June 2020 when all in-person clinical research halted at our institution due to COVID, and after completion of the interim analysis, enrollment was permanently halted in August 2022.
Pre-assignment Details: Altogether, 1823 patients were screened and 209 were randomized into the study.
Period: Overall Study
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
Started | 104 | 105
Completed | 102 | 102
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg | Total
Number analyzed (Participants) | 104 | 105 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11) | 37 (11) | 38.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 83 | 179
  Male | 8 | 22 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 104 | 105 | 209
Duration of Headache [Median (Inter-Quartile Range); unit: hours] | 48 [12 to 96] | 48 [15 to 72] | 48 [12 to 96]
Aura Symptoms [Count of Participants; unit: Participants]
  No | 62 | 64 | 126
  Yes | 42 | 41 | 83
Treated Migraine Before Heading to the Emergency Department (ED) [Count of Participants; unit: Participants]
  No | 35 | 42 | 77
  Yes | 69 | 63 | 132
Headache Intensity [Count of Participants; unit: Participants]
  Moderate | 27 | 31 | 58
  Severe | 77 | 74 | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Headaches Who Have Sustained Headache Relief for 48 Hours
Description: The number of subjects achieving sustained headache relief for 48 hours and maintaining this level, without requiring additional rescue therapy for the entire 48 hour follow up period, will be determined. Headache relief will be defined as the number of subjects reporting a headache intensity of either "none" or "mild."
Time Frame: 48 hours
Population: Two subjects in the Dexamethasone 4mg arm and 3 subjects in the Dexamethasone 16mg arm did not complete their 48 hour follow up. As such, 48 hour data was not collected from these subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
Number analyzed (Participants) | 102 | 102
Participants | 35 | 42
Statistical Analysis 1: Comparison: Dexamethasone 4mg vs Dexamethasone 16mg; Test type: Superiority; Risk Ratio (RR) = 7, 95% CI 2-sided [-6 to 20]

2. Secondary Outcome: Number of Subjects With Headache Who Have Relief Within Two Hours of Medication Administration
Description: The number of subjects who achieve a headache intensity level of either "none" or "mild" within two hours of medication administration, without requiring rescue medication, will be determined.
Time Frame: Two hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
Number analyzed (Participants) | 104 | 105
Participants | 77 | 82
Statistical Analysis 1: Comparison: Dexamethasone 4mg vs Dexamethasone 16mg; Test type: Superiority; Risk Ratio (RR) = 4, 95% CI 2-sided [-8 to 16]

3. Secondary Outcome: Additional Headache Medication in the ED
Description: The number of participants requiring the use of additional headache medication (rescue therapy) during their time in the ED will be determined.
Time Frame: Up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
Number analyzed (Participants) | 104 | 105
Participants
  No | 83 | 87
  Yes | 21 | 18
Statistical Analysis 1: Comparison: Dexamethasone 4mg vs Dexamethasone 16mg; Test type: Superiority; Risk Ratio (RR) = 3, 95% CI 2-sided [-8 to 14]

4. Secondary Outcome: Patient Preference for Receiving the Same Medication for a Subsequent Headache
Description: During the 48 hour follow up patients were queried as to whether they would want the same headache treatment regimen during the onset of a subsequent headache. The number of responses were tabulated and reported.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
Number analyzed (Participants) | 102 | 102
Participants
  Yes | 80 | 83
  No | 12 | 7
  Not sure | 10 | 12

5. Secondary Outcome: Number of Days With Headache
Description: The median number of headache days during the week after ED discharge will be determined.
Time Frame: One week
Population: Two subjects in the Dexamethasone 4mg arm and 3 subjects in the Dexamethasone 16mg arm were lost to follow up. Data was not collected from these subjects.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
Number analyzed (Participants) | 102 | 102
days | 2 [1 to 5] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Dexamethasone 4mg vs Dexamethasone 16mg; Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.3 to 1.2]

6. Secondary Outcome: Use of Additional Headache Medication After ED Discharge
Description: The number of participants requiring the use of additional headache medication following ED discharge will be summarized.
Time Frame: Up to 24 hours
Population: Data related to additional headache medication is missing for 4 participants in each treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
Number analyzed (Participants) | 100 | 101
Participants
  No | 55 | 60
  Yes | 45 | 41
Statistical Analysis 1: Comparison: Dexamethasone 4mg vs Dexamethasone 16mg; Test type: Superiority; Risk Ratio (RR) = 4, 95% CI 2-sided [-9 to 18]

ADVERSE EVENTS:
Time Frame: Up to 48 hours
Arm/Group | Dexamethasone 4mg | Dexamethasone 16mg
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/105
Serious Adverse Events (participants affected / at risk) | 2/104 | 0/105
Other Adverse Events (participants affected / at risk) | 22/104 | 24/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone 4mg (N=104) | Dexamethasone 16mg (N=105)
Cerebellar Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Verbatim Term: Markedly Elevated Blood Sugar
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone 4mg (N=104) | Dexamethasone 16mg (N=105)
Somnolence (Nervous system disorders) | 4 | 9 — Verbatim Term: Drowsiness
Dizziness (Nervous system disorders) | 5 | 4
Akathisia (Nervous system disorders) | 8 | 7
Fatigue (General disorders) | 3 | 2 — Verbatim Terms: Weakness, Lack of Energy
Stomach Pain (Gastrointestinal disorders) | 2 | 1 — Verbatim Term: Stomach ache
Palpitations (Cardiac disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT04112823/Prot_SAP_000.pdf